CLINICAL TRIAL: NCT02708706
Title: The Efficacy of Ultrasound-guided Hydrodilatation With Hyaluronic Acid for Patients With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-10-009B
Record Dates: First submitted 2016-02-15; First posted 2016-03-15 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; hyaluronic acid
MeSH Terms: conditions — Bursitis | interventions — Hyaluronic Acid; Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- physical therapy and hyaluronic acid (Experimental): patient received ultrasound-guided hydrodilatation with hyaluronic acid plus physical therapy
  Interventions: Drug: hyaluronic acid (hyruan); Other: physical therapy
- physical therapy only (Active Comparator): patient received physical therapy only
  Interventions: Other: physical therapy

INTERVENTIONS:
Drug: hyaluronic acid (hyruan) — 2cc hyaluronic acid
  Other Names: hyaluronate
  Arms: physical therapy and hyaluronic acid
Other: physical therapy — patient received traditional physical therapy, including therapeutic exercise and stretch exercise
  Other Names: rehabilitation

SUMMARY:
This study was conducted to compare the efficacy of hydrodilatation with hyaluronic acid under ultrasonographic guidance plus physical therapy (PT) with that of PT alone for treating adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis is a common cause of shoulder pain, and the efficacy of most interventions is limited. This study was conducted to compare the efficacy of hydrodilatation with hyaluronic acid under ultrasonographic guidance plus physical therapy (PT) with that of PT alone for treating adhesive capsulitis.

Design: a prospective, single-blinded, randomized, clinical trial

Patient and methods:

Patients with adhesive capsulitis for at least 3 months were enrolled and randomly allocated into group 1 (hydrodilatation with hyaluronic acid under ultrasonographic guidance plus PT) and group 2 (PT alone). The patients were evaluated before treatment and were reevaluated 0, 6, and 12 weeks after the beginning of the treatment. Outcomes measures included a pain scale (visual analog scale), range of motion, Constant shoulder score, Shoulder Pain And Disability Index, and the Short Form-36

ELIGIBILITY:
Inclusion Criteria:

1. a duration of complaints more than 3 months
2. a reduction in passive range of motion in at least 2 of the following: forward flexion, abduction, or external rotation of the affected shoulder of more than 30 degree compared with the other side.

Exclusion Criteria:

1. prior manipulation of the affected shoulder under anesthesia;
2. other conditions involving the shoulder ( rheumatoid arthritis, Hill-Sachs lesions, osteoarthritis, damage to the glenohumeral cartilage,osteoporosis, or malignancies in the shoulder region);
3. neurologic deficits affecting shoulder function in normal daily activities;
4. shoulder pain caused by cervical radiculopathy
5. a history of drug allergy to hyaluronic acid;
6. pregnancy or lactation;
7. received injection into the affected shoulder during the preceding 3 months

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
change in constant shoulder score | at 6, 12 wk
  visual analog scale

SECONDARY OUTCOMES:
change in glenohumeral joint range of motion | at 6, 12 wk
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position.
change in Short Form-36 | at 6, 12 wk
  The SF-36 consists of eight sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
change in pain intensity | at 6, 12 wk
  pain intensity was measured by visual analog scale.
change in Shoulder Pain And disability index | at 6, 12 wk
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei veteran general hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu SY, Hsu PC, Tsai YY, Huang JR, Wang KA, Wang JC. Efficacy of combined ultrasound-guided hydrodilatation with hyaluronic acid and physical therapy in patients with adhesive capsulitis: A randomised controlled trial. Clin Rehabil. 2024 Feb;38(2):202-215. doi: 10.1177/02692155231200089. Epub 2023 Sep 11. PMID 37697666